CLINICAL TRIAL: NCT06722313
Title: Optimized PGT-M Strategy Using Gametes or Arrested Embryos from Patients with No Proband
Brief Title: Optimized PGT-M Strategy for Patients with No Proband
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JIAI E2023-12
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: De Novo Mutation; Preimplantation Genetic Testing; Without Proband
Keywords: preimplantation genetic testing; without proband; De Novo Mutation
MeSH Terms: interventions — Sperm Count; Biopsy; Vitrification; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PGT-M (Experimental): The couples intended for PGT-M without proband were recruited from Shanghai JiAi Genetics and IVF Institute, Obstetrics and Gynecology Hospital of Fudan University between January 2023 and December 2024, and were included in the study if they were expected to have difficulties in the identification of an embryo as proband.
  Interventions: Diagnostic Test: Gametes (sperm or second polar bodies, MI eggs) or arrested embryos were reserved for identification of a proband

INTERVENTIONS:
Diagnostic Test: Gametes (sperm or second polar bodies, MI eggs) or arrested embryos were reserved for identification of a proband — 1. Targeted deep sequencing for mosaicism detection for patients with suspected gonadal mosaicism, eg. Repeated similar abortion due to the same variant while the couple were tested negative for the variant in the peripheral blood.
  2. Ovarian stimulation, embryo culture, biopsy and vitrification as routinely used in the IVF clinical practice.
  3. Gametes and arrested embryo preservation by the embryo laboratory during embryo culture.
  4. Genetic testing, including multiple displacement amplification for WGA, variant sequencing in WGA products and Infinium Chip protocol for amplified DNA and haplotype analysis
  Other Names: Targeted deep sequencing for mosaicism detection; Ovarian stimulation, embryo culture, biopsy and vitrification; Genetic testing

SUMMARY:
The clinical practice of PGT-M for monogenetic disease usually adopted a double-checking strategy, which detect the mutation by Sanger sequencing and meantime construct haplotypes using the DNA sample of the proband so as to avoid the risks of misdiagnosis due to recombination and allele drop out (ADO). When there is no affected parent or offspring to serve as the proband, embryo carriers identified through direct mutation detection can be preferentially taken as probands for subsequent linkage analysis. In cases where none of the embryos are detected as mutant carrier, single sperm or the second polar body (PB2) can be complementally collected in the work-up of haplotype establishment. Our study aims to develop an optimized strategy of haplotype construction using gametes or arrested embryos for PGT-M in pedigrees with single gene diseases and no proband in the setting of difficult cases, which takes into account the expected number of oocytes acquired and the gonadal mosaicism.

ELIGIBILITY:
Inclusion Criteria:

* The couples intended for PGT-M without proband were recruited from Shanghai JiAi Genetics and IVF Institute, Obstetrics and Gynecology Hospital of Fudan University between January 2023 and December 2024, and were included in the study if they were expected to have difficulties in the identification of an EAP, typically meeting one of the following criteria:

  1. the carrier of the pathogenic variant was without typical clinical symptoms or detected as gonadosomal mosaic;
  2. the asymptomatic parents, who had one or more children affected with the same disorder, did not possess the genomic alterations carried by the children as per Sanger sequencing or targeted deep sequencing;
  3. female partner with diminished ovarian reserve and therefore a low yield of embryos;
  4. the variants are X-linked and the karyotype of the variant carrier is 47, XXX or 47, XXY etc.

Exclusion Criteria:

* (1) Non-PGT-M families; (2) Pedigree of other proband samples can be obtained; (3) Patients seeking for PGT-M who strongly request no haplotype analysis in embryos and only require Sanger testing after being fully informed of the risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Consistence of the PGT-M with prenatal diagnosis with amniocentesis | 16 weeks of gestation
  whether the PGT-M result of the embryos are consistent with the prenatal genetic testing result of amniocentesis

CONTACTS AND LOCATIONS:
Overall Officials: Yilun Sui, MD, Principal Investigator — Shanghai Ji Ai Genetics and IVF Institute, Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Shanghai Ji Ai Genetics and IVF Institute, Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The de-identified IPD will be published along with the publications of this study
Supporting Information: Study Protocol

REFERENCES:
- [Background] Summerer A, Schafer E, Mautner VF, Messiaen L, Cooper DN, Kehrer-Sawatzki H. Ultra-deep amplicon sequencing indicates absence of low-grade mosaicism with normal cells in patients with type-1 NF1 deletions. Hum Genet. 2019 Jan;138(1):73-81. doi: 10.1007/s00439-018-1961-5. Epub 2018 Nov 26. PMID 30478644
- [Background] Xiao M, Shi H, Rao J, Xi Y, Zhang S, Wu J, Zhu S, Zhou J, Xu H, Lei C, Sun X. Combined Preimplantation Genetic Testing for Genetic Kidney Disease: Genetic Risk Identification, Assisted Reproductive Cycle, and Pregnancy Outcome Analysis. Front Med (Lausanne). 2022 Jun 17;9:936578. doi: 10.3389/fmed.2022.936578. eCollection 2022. PMID 35783601
- [Background] Wilde AAM, Amin AS. Clinical Spectrum of SCN5A Mutations: Long QT Syndrome, Brugada Syndrome, and Cardiomyopathy. JACC Clin Electrophysiol. 2018 May;4(5):569-579. doi: 10.1016/j.jacep.2018.03.006. Epub 2018 May 2. PMID 29798782
- [Background] Wang Y, Zhai F, Guan S, Yan Z, Zhu X, Kuo Y, Wang N, Zhi X, Lian Y, Huang J, Jia J, Liu P, Li R, Qiao J, Yan L. A comprehensive PGT-M strategy for ADPKD patients with de novo PKD1 mutations using affected embryo or gametes as proband. J Assist Reprod Genet. 2021 Sep;38(9):2425-2434. doi: 10.1007/s10815-021-02188-z. Epub 2021 May 3. PMID 33939064